CLINICAL TRIAL: NCT01506596
Title: A Phase II Study of Pazopanib in the Treatment of Surgically Unresectable or Metastatic Liposarcoma
Brief Title: Study of Pazopanib in the Treatment of Surgically Unresectable or Metastatic Liposarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vector Oncology (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABLSMLS1101
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-03

CONDITIONS: Liposarcoma; Surgically Unresectable Liposarcoma; Metastatic Liposarcoma
Keywords: Liposarcoma
MeSH Terms: conditions — Liposarcoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pazopanib (Experimental): Pazopanib 800 mg orally once daily will be started on Cycle 1 Day 1 and will be administered continuously for a 28-day cycle. Study treatment may continue until disease progression or unacceptable toxicity.
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — Pazopanib 800 mg orally once daily will be started on Cycle 1 Day 1 and will be administered continuously for a 28-day cycle. Study treatment may continue until disease progression or unacceptable toxicity.
  Other Names: Votrient

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of single agent pazopanib in subjects with unresectable or metastatic liposarcoma.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, prospective, open label, single arm study. The primary endpoint of the study is progression-free rate as defined by Response Evaluation Criteria in Solid Tumors (RECIST) guidelines version 1.1 at week 12 after start of treatment. The secondary endpoints include overall progression-free survival (PFS), response rate (RR), duration of response, overall survival (OS), and toxicity assessment through the reporting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age > or = to 18 years.
* Histologically or cytologically confirmed high- or intermediate-grade liposarcoma (allowed subtypes include liposarcoma dedifferentiated, myxoid/round cell, pleomorphic, mixed-type, or not otherwise specified).
* Surgically unresectable or metastatic disease.
* Any number of prior treatment treatment regimens, including treatment naive subjects.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Measurable or evaluable (non-measurable) disease per RECIST guidelines version 1.1. Subjects must have documented disease progression within the past 6 months.
* Adequate organ system function determined within 14 days prior to first dose of study treatment.
* Left ventricular ejection fraction (LVEF) > 50% of the institutional LLN within 28 days prior to the first dose of study treatment.
* Females must be of either non-child bearing potential or have a negative pregnancy test within 7 days prior to the first dose of study treatment.

Exclusion Criteria:

* Well differentiated liposarcoma.
* Prior treatment with tyrosine kinase inhibitors (TKIs) or vascular endothelial growth factor (VEGF) inhibitors.
* Prior malignancy (Note: subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible).
* History or clinical evidence of central nervous system metastases or leptomeningeal carcinomatosis, unless previously treated, asymptomatic, and off steroids and anti-seizure medication for 6 months prior to first dose of study drug
* Clinically significant gastrointestinal (GI) abnormalities that may increase the risk for GI bleeding.
* Clinically significant GI abnormalities that may affect absorption of investigational product.
* Presence of uncontrolled infection.
* Corrected QT interval > 480 msecs using Bazett's formula.
* History of certain cardiovascular conditions within the past 6 months.
* Poorly controlled hypertension [defined as systolic blood pressure of > or = 140 mmHg or diastolic blood pressure > or = 90 mmHg].
* History of cerebrovascular accident including transient ischemic attack, pulmonary embolism, or untreated deep vein thrombosis within the past 6 months.
* Prior major surgery or trauma within 28 days prior to the first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.
* Hemoptysis in excess of 2.5 mL within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug, whichever is longer, prior to the first dose of study drug and for the duration of study treatment.
* Radiation therapy, minor surgery, tumor embolization, chemotherapy, immunotherapy, biologic therapy, investigational therapy, or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug.
* Administration of any non-oncologic investigational drug within 30 days or five half-lives (whichever is longer) prior to receiving the first dose of study drug.
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.
* Known immediate or delayed hypersensitivity reaction to idiosyncrasy to drugs chemically realted to pazopanib or excipients that contraindicates participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03; Primary Completion 2014-10 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Samuels, MD, Study Chair — Northwest Oncology
Locations (9):
- United States (9):
  - Sarcoma Oncology Center, Santa Monica, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Kootenai Cancer Center, Post Falls, Idaho
  - Oncology Specialists, SC, Niles, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - West Clinic, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pazopanib
Started | 42
Completed | 41 (One enrolled patient had ineligible pathology after starting treatment; was removed from treatment.)
Not Completed | 1
Not completed — ineligible pathology | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (15.52)
Gender [Count of Participants; unit: Participants]
  Female | 14
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: 12-week Progression Free Rate
Description: Progression will be as defined per Response Evaluation Criteria In Solid Tumors (RECIST) guidelines version 1.1. Subjects who remain under observation and progression free at 12 weeks will be defined as treatment successes. Subjects who progress per RECIST by 12 weeks or who drop out without evidence of progression prior to 12 weeks will be defined as treatment failures.Progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST v1.1), as a >=20% increase in the sum of diameters of target lesions, or a measurable increase in a non-target lesion, or the appearance of >=1 new lesion.
Time Frame: Assessed after 12 weeks of study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 41
percentage of participants | 68.29 [51.91 to 81.92]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was measured from date of consent until the subject experiences disease progression (assessed approximately every 12 weeks) or death, whichever came first, up to 27 months. Repeat radiologic imaging will be conducted after every 3 cycles of treatment (approximately every 12 weeks) to evaluate disease status per RECIST v1.1. Subjects who discontinue study treatment for reasons other than disease progression will continue to have their disease status reported every 3 months post end of treatment up to 27 months.
Time Frame: Date of Consent until progression or death, up to 27 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 41
months | 4.44 [3.2 to 6.5]

3. Secondary Outcome: Best Overall Response
Description: Best overall response is defined as the best response across all time points. Repeat radiologic imaging was conducted after every 3 cycles of treatment (approximately every 12 weeks). Response was evaluated using RECIST v1.1 guidelines, where complete response (CR) is the disappearance of all target and non-target lesions; partial response (PR) is >=30% decrease in the sum of diameters of target lesions; progressive disease (PD) is >=20% increase in the sum of diameters of target lesions, or a measurable increase in a non-target lesion, or the appearance of >=1 new lesion; stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: Date of consent until end of study treatment, up to 32 months
Measure: Number; unit: percentage of participants
Arm/Group | Pazopanib
Number analyzed (Participants) | 41
percentage of participants
  Complete response | 0
  Partial Response | 2.4
  Stable Disease | 41.5
  Progressive Disease | 43.9
  Inevaluable | 12.2

4. Secondary Outcome: Duration of Response
Description: Response is defined as Complete Response (CR) or Partial Response (PR) per RECIST v1.1. Repeat radiologic imaging will be conducted after every 3 cycles of treatment (approximately every 12 weeks) to evaluate disease status per RECIST v1.1. Confirmation of CR or PR is required by repeat scans that should be performed 4 weeks after the criteria for response are first met.
Time Frame: Measure of the amount of time that the criteria for response per RECIST are first met until disease progression
Population: Since so few patients experienced a response, the pre-specified endpoint of duration of response was not analyzed.
Arm/Group | Pazopanib
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from date of consent until time of death from any cause, up to 32 months.
Time Frame: Date of Consent until death, up to 32 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib
Number analyzed (Participants) | 41
months | 12.62 [8.5 to 16.2]

ADVERSE EVENTS:
Arm/Group | Pazopanib
Serious Adverse Events (participants affected / at risk) | 17/41
Other Adverse Events (participants affected / at risk) | 39/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=41)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Gastric Perforation (Gastrointestinal disorders) | 2
Large Intestine Perforation (Gastrointestinal disorders) | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
death (General disorders) | 2
Fatigue (General disorders) | 1
Hepatic Haemorrhage (Hepatobiliary disorders) | 1
Cellulitis (Infections and infestations) | 1
Escherichia Sepsis (Infections and infestations) | 1
Perirectal Abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
International Normalised Ratio Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depressed Level Of Consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Transient Ischaemic Attack (Nervous system disorders) | 1
Mental Disorder Due To A General Medical Condition (Psychiatric disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Pazopanib (N=41)
Anaemia (Blood and lymphatic system disorders) | 7
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 8
Exfoliation Syndrome (Eye disorders) | 1
Exophthalmos (Eye disorders) | 1
Eye Swelling (Eye disorders) | 1
Periorbital Oedema (Eye disorders) | 1
Scleral Disorder (Eye disorders) | 2
Vision Blurred (Eye disorders) | 2
Abdominal Distension (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 9
Abdominal Pain Lower (Gastrointestinal disorders) | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 4
Colonic Fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Dental Caries (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 14
Dry Mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Gastrointestinal Fistula (Gastrointestinal disorders) | 1
Gastrointestinal Motility Disorder (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 1
Large Intestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Proctalgia (Gastrointestinal disorders) | 2
Proctitis (Gastrointestinal disorders) | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 3
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 1
Chest Pain (General disorders) | 1
Early Satiety (General disorders) | 1
Fatigue (General disorders) | 12
Localised Oedema (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Oedema Peripheral (General disorders) | 5
Pain (General disorders) | 1
Peripheral Swelling (General disorders) | 2
Pyrexia (General disorders) | 1
Temperature Intolerance (General disorders) | 1
Diverticulitis (Infections and infestations) | 1
Gastrointestinal Infection (Infections and infestations) | 1
Herpes Zoster (Infections and infestations) | 1
Nail Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 4
Fall (Injury, poisoning and procedural complications) | 2
Stress Fracture (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
Transfusion Reaction (Injury, poisoning and procedural complications) | 1
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Alanine Aminotransferase Increased (Investigations) | 3
Aspartate Aminotransferase Increased (Investigations) | 2
Blood Bilirubin Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 4
Blood Culture Positive (Investigations) | 1
Blood Thyroid Stimulating Hormone Increased (Investigations) | 2
Electrocardiogram QT Prolonged (Investigations) | 1
Gastrointestinal Infection (Investigations) | 1
International Normalised Ratio Increased (Investigations) | 1
Lipase Increased (Investigations) | 1
Neutrophil Count Decreased (Investigations) | 2
Platelet Count Decreased (Investigations) | 7
Prothrombin Time Prolonged (Investigations) | 1
Troponin I Increased (Investigations) | 1
Urine Output Decreased (Investigations) | 1
Urine Protein/Creatinine Ratio (Investigations) | 3
Weight Decreased (Investigations) | 7
Decreased Appetite (Metabolism and nutrition disorders) | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Iron Deficiency (Metabolism and nutrition disorders) | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 4
Fistula (Musculoskeletal and connective tissue disorders) | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Salivary Gland Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Disturbance In Attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 7
Dysgeusia (Nervous system disorders) | 6
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Metabolic Encephalopathy (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Vocal Cord Paralysis (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusional State (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Restlessness (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Testicular Swelling (Reproductive system and breast disorders) | 1
Vaginal Haemorrhage*f (Reproductive system and breast disorders) | 1/14 — *f: Adverse Event was female specified, and percentage was based on female population(Nf=14).
Vulvovaginal Dryness*f (Reproductive system and breast disorders) | 2/14 — *f: Adverse Event was female specified, and percentage was based on female population(Nf=14).
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 2
Granulomatous Dermatitis (Skin and subcutaneous tissue disorders) | 1
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 3
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Nail Discolouration (Skin and subcutaneous tissue disorders) | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Rash Macular (Skin and subcutaneous tissue disorders) | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 2
Skin Exfoliation*m (Skin and subcutaneous tissue disorders) | 1/27 — *m: Adverse Event was male specified, and percentage was based on male population(Nm=27).
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Skin Mass (Skin and subcutaneous tissue disorders) | 1
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 3
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 15
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution/PI may use Institution/PI derived Study results in a Publication provided Publication does not disclose Vector Confidential Information unnecessary to publish Study results. Institution/PI will submit to Vector for review/comment proposed Publication and data necessary for meaningful review at least 30 days prior to submission. Vector may request delay of submission up to 60 days in order to file patent applications relating to an Invention.